CLINICAL TRIAL: NCT03431168
Title: The PREMISE Trial: A Novel Regimen to Prevent Malaria and Sexually Transmitted Infections in Pregnant Women With HIV
Brief Title: A Novel Regimen to Prevent Malaria and STI in Pregnant Women With HIV
Acronym: PREMISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jodie A. Dionne, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-300001112
Record Dates: First submitted 2018-01-02; First posted 2018-02-13 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: HIV; Pregnancy Malaria; Sexually Transmitted Infection
Keywords: STI Prevention; Cameroon; sub-Saharan Africa; HIV pregnancy; Malaria in pregnancy
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azithromycin/TMPS (Active Comparator): Azithromycin 1 gm po daily x 3 days at enrollment and at each 4 week follow up visit.
  TMPS double strength 1 tablet po daily.
  Interventions: Drug: Azithromycin/TMPS
- Placebo/TMPS (Placebo Comparator): Azithromycin placebo 1 gm po daily x 3 days at enrollment and at each 4 week follow up visit.
  TMPS double strength 1 tablet po daily.
  Interventions: Drug: Placebo/TMPS

INTERVENTIONS:
Drug: Azithromycin/TMPS — 2 tabs po daily x 3 days at enrollment and at each monthly follow up visit
  Other Names: Cotrimoxazole
  Arms: Azithromycin/TMPS
Drug: Placebo/TMPS — 2 tabs po daily x 3 days at enrollment and at each monthly follow up visit
  Other Names: Co-Trimoxazole
  Arms: Placebo/TMPS

SUMMARY:
More than 3 billion people worldwide are at risk of acquiring malaria and pregnant women living with HIV in Africa are at particular risk. An effective prophylaxis regimen capable of preventing malaria and other common perinatal infections would have great potential to improve adverse birth outcomes. The purpose of this randomized controlled trial is to evaluate a new combination prophylaxis regimen in pregnant women with HIV in Cameroon to determine its efficacy and safety.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends malaria prophylaxis for all pregnant women living in endemic areas in order to reduce maternal anemia, low birth weight and perinatal mortality by 25-45%. The most commonly used regimen is intermittently dosed sulfadoxine-pyrimethamine (SP).Unfortunately, SP prophylaxis is contraindicated for HIV-infected pregnant women since co-administration with TMPS (trimethoprim-sulfamethoxazole) causes serious adverse events. TMPS (Bactrim or Cotrimoxazole) is an effective, well-tolerated, low-cost antibiotic that is used as prophylaxis in HIV-patients with low CD4 counts. It has anti-malarial activity with prophylactic efficacy that is comparable to SP (30-90%). Daily TMPS is recommended as malaria prophylaxis in pregnant women with HIV in many African countries (including Cameroon) but malaria infection rates are high even when medication compliance is excellent; thus, new and improved options are urgently needed. Azithromycin (AZ) is a macrolide antibiotic with activity against malaria, a good safety profile in pregnancy and proven utility as a part of combination malaria prevention regimens (such as SP-AZ). It also has activity against sexually transmitted infections (STI) and perinatal pathogens, including chlamydia (CT), gonorrhea (GC), syphilis and GBS (Streptococcus agalactiae or Group B Streptococcus), a potential but understudied contributor to high rates of newborn sepsis and death in Africa. SP-AZ prophylaxis in HIV-uninfected pregnant women has been reported to reduce prevalence of low birth weight (RR 0.74, 95% confidence interval (CI) 0.6-0.9) and preterm delivery (RR 0.66, 95% CI 0.48-0.91) compared to SP alone.

Thus, the central hypothesis is that a TMPS-AZ combination will be more effective than standard TMPS malaria prophylaxis in pregnant women with HIV, and that it will also decrease STI coinfection. Investigators plan a test-of-concept of the central hypothesis by conducting a double blinded, Phase II randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-infection (documented in medical record)
* Age ≥16 years
* Confirmed pregnancy, <28 weeks estimated gestational age (by best obstetric estimate which may include ultrasound or fundal height and LMP)
* Live singleton pregnancy
* Receiving prenatal care at Mboppi Hospital or Mutengene Hospital
* Plan to receive follow up prenatal care and deliver at study facility
* Capable of providing written informed consent
* Able and agree to come to facility for febrile episodes or acute illness during pregnancy (with reimbursement of transportation costs).
* Agree to avoid antimalarial medications outside of study protocol.

Exclusion Criteria:

* Severe anemia (last hemoglobin <6)
* History of severe adverse reaction to co-trimoxazole or azithromycin
* Active medical problem requiring inpatient evaluation at the time of screening
* Intention of moving far away from the facility during pregnancy or not likely to return for follow up care or delivery
* Signs or symptoms of early or active labor
* History of severe cardiac disease (including congestive heart failure, severe valvular disease or arrhythmias).

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 308 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jodie A Dionne-Odom, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin/TMPS: Azithromycin 1 gm po daily x 3 days at enrollment and at each 4 week follow up visit.
  TMPS double strength 1 tablet po daily.
  Azithromycin/TMPS: 2 tabs po daily x 3 days at enrollment and at each monthly follow up visit
- Placebo/TMPS: Azithromycin placebo 1 gm po daily x 3 days at enrollment and at each 4 week follow up visit.
  TMPS double strength 1 tablet po daily.
  Placebo/TMPS: 2 tabs po daily x 3 days at enrollment and at each monthly follow up visit
Period: Overall Study
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Started | 155 | 153
Completed | 132 | 129
Not Completed | 23 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin/TMPS | Placebo/TMPS | Total
Number analyzed (Participants) | 155 | 153 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 153 | 308
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 36] | 32 [28 to 36] | 32 [28 to 36]
Sex: Female, Male [Count of Participants; unit: Participants] — All pregnant females
  Participants
    Female | 155 | 153 | 308
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 155 | 153 | 308
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Cameroon
  participants
    Cameroon | 155 | 153 | 308

OUTCOME MEASURES:

1. Primary Outcome: Plasmodium Falciparum Peripheral Parasitemia
Description: P. falciparum detected by microscopy or polymerase chain reaction (PCR)
Time Frame: At end of pregnancy (>35 weeks) or at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 140 | 136
Participants | 8 | 7

2. Primary Outcome: Proportion With Composite STI Outcome
Description: Including chlamydia (NAAT (nucleic acid amplification test) positive) , gonorrhea (NAAT positive), syphilis (non-treponemal and treponemal test positive) infections.
Time Frame: will be measured in both groups (>35 weeks) or at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 140 | 133
Participants | 2 | 2

3. Secondary Outcome: Low Birthweight (<2500 Grams)
Description: Neonatal weight measured with digital scale
Time Frame: at birth
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 141 | 137
Participants | 4 | 7

4. Secondary Outcome: Proportion With Adverse Birth Outcomes
Description: Composite measure: low infant birthweight (<2500 grams), miscarriage (<28 weeks), preterm delivery (<37 weeks), small for gestational age (SGA), congenital anomaly detected on surface examination, early neonatal mortality (within 7 days of birth)
Time Frame: Birth outcomes will be measured at birth for all outcomes except early neonatal mortality defined as within 7 days of birth. Early neonatal mortality will be assessed at a six week follow up phone call.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 155 | 153
Participants | 13 | 20

5. Secondary Outcome: Maternal Adherence to the Prophylactic Regimen
Description: Directly observed therapy (DOT) in clinic for the 1st dose of study medication. Self-report and pill count will be used to assess adherence and maternal tolerability for study medications taken at home from the time of enrollment until delivery. At each follow up visit and at delivery, participants will complete a medication adherence survey. They will self-report adherence to the 3 day study regimen (AZ or placebo).
Time Frame: Adherence of study medication taken at home will be documented from the date of randomization until the time of delivery, assessed up to 42 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 148 | 148
Participants | 148 | 148

6. Secondary Outcome: Proportion of Participants With Symptomatic Malaria
Description: Fever and positive malaria test (rapid diagnostic test) at routine visits or sick call visits or maternal report of malaria diagnosis.
Time Frame: From the date of randomization until the time of delivery, assessed up to 42 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 148 | 148
Participants | 13 | 13

7. Secondary Outcome: Proportion With Placental Malaria
Description: Placentas will be collected on a subset of women and impression smear will be used to assess for malaria infection
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 35 | 35
Participants | 7 | 5

8. Secondary Outcome: Proportion With Maternal Anemia and Severe Maternal Anemia
Description: anemia defined as hemoglobin <11 g/dL, severe anemia defined as hemoglobin <7 g/dL.
Time Frame: At the end of pregnancy (>35 weeks) or at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 148 | 148
Participants | 2 | 2

9. Secondary Outcome: Composite STI Measure (Including All STI Tests)
Description: Proportion of women with GC/CT (by NAAT), syphilis (by serology), Mycoplasma genitalium (NAAT).
Time Frame: After 35 weeks GA or at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 155 | 153
Participants | 5 | 5

10. Secondary Outcome: GBS Colonization
Description: anogenital GBS colonization detected by NAAT (PCR)
Time Frame: at or near term or at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
Number analyzed (Participants) | 147 | 144
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: From enrollment during the 2nd trimester through delivery
Arm/Group | Azithromycin/TMPS | Placebo/TMPS
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/153
Other Adverse Events (participants affected / at risk) | 0/155 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03431168/Prot_SAP_ICF_000.pdf